CLINICAL TRIAL: NCT05707676
Title: A Phase I，Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of LB4330 in Patients With Advanced Solid Tumors（MEETCD8-001）
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of LB4330 in Patients With Advanced Solid Tumors（MEETCD8-001）
Acronym: MEETCD8-001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to adjustments in the sponsor's development strategy, it has been decided to terminate the study.
Sponsor: L & L Bio Co., Ltd., Ningbo, China (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB4330-CHN-I-01
Record Dates: First submitted 2022-12-28; First posted 2023-02-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: LB4330

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Dose escalation uses an accelerated titration design combined with the standard 3+3 method.The planned maximum sample size for the dose-escalation phase is 39 subjects, with a maximum of 6 subjects per dose level.
  Interventions: Drug: LB4330
- Single Drug Expansion (Experimental): Planned cohorts and subject numbers:Cohort A: Advanced gastric and gastroesophageal junction adenocarcinoma with Claudin 18.2 expression that has failed standard treatment, with no more than three prior lines of therapy (up to 15 patients); Cohort B: Advanced pancreatic ductal adenocarcinoma with Claudin 18.2 expression that has failed standard treatment, with no more than three prior lines of therapy (up to 30 patients); Cohort C: Other advanced solid tumors with Claudin 18.2 expression that have failed standard treatment, with no more than three prior lines of therapy (a total of up to 15 patients); Cohort D: Advanced solid tumors without Claudin 18.2 expression (limited to ovarian cancer, cholangiocarcinoma, pancreatic cancer, gastric and gastroesophageal junction cancer) that have failed treatment, with no more than three prior lines of therapy (a total of up to 20 patients).
  Interventions: Drug: LB4330

INTERVENTIONS:
Drug: LB4330 — LB4330

SUMMARY:
This is a Phase I study designed to evaluate if LB4330, an anti-Claudin 18.2 and CD8 T cell activator fusion protein, is safe, tolerable and efficacious in participants with Advanced Solid Tumors

DETAILED DESCRIPTION:
This first time in patients, open-label, multi-center study will have LB4330 administered intravenously (IV) in Patients with Advanced Solid Tumors. This study will have 2 parts: Part A which will have dose escalation cohorts and Part B which will have the dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be eligible for enrollment:

1. Age between 18 and 75 years (inclusive), regardless of sex. 2.

* Dose-Escalation Phase: Histologically or cytologically confirmed advanced malignant solid tumors.
* Monotherapy Expansion Phase: Histologically or cytologically confirmed advanced gastric/gastroesophageal junction adenocarcinoma, pancreatic ductal adenocarcinoma, or other solid tumors that have failed standard treatment, or for which there is no standard treatment, or for whom standard treatment is currently unsuitable. 3.
* Dose-Escalation Phase: At least one evaluable lesion based on RECIST v1.1.
* Monotherapy Expansion Phase: At least one measurable lesion based on RECIST v1.1 (lesions previously treated with radiotherapy or localized therapy are not considered measurable unless they have clearly progressed or persisted for at least 3 months post-radiotherapy).
* Monotherapy Expansion Phase: Must provide a prior Claudin 18.2 test report; if unavailable, archived or fresh tumor tissue samples must be submitted.
* Cohort E: If Claudin 18.2 testing has been done previously, the result must show no Claudin 18.2 expression. If no test result is available and no sample can be provided, inclusion is allowed upon joint agreement between the sponsor and investigator.
* Cohorts A, B, C: Require Claudin 18.2 expression (≥1% of tumor cells with staining intensity of 1+ or above).
* Cohort D: Must be Claudin 18.2 negative.
* Cohort E: Must not have known Claudin 18.2 expression (≥1% of tumor cells with staining intensity of 1+ or above).

  5. ECOG performance status of 0-1. 6. Expected survival time of at least 3 months. 7. Adequate organ function:

Hematologic (no transfusion or hematopoietic growth factors within 14 days prior):

* ANC ≥ 1.5 × 10⁹/L
* Platelets ≥ 100 × 10⁹/L
* Hemoglobin ≥ 90 g/L

Liver Function:

* Total bilirubin (TBIL) ≤ 1.5 × ULN; ≤ 3 × ULN if hepatic metastases or Gilbert's syndrome present
* ALT ≤ 3 × ULN (≤ 5 × ULN for liver metastases or HCC)
* AST ≤ 3 × ULN (≤ 5 × ULN for liver metastases or HCC)

Renal Function:

* Serum creatinine ≤ 1.5 × ULN
* Creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula)

Coagulation:

* APTT ≤ 1.5 × ULN
* INR ≤ 1.5 × ULN 8. Fertile patients (male and female) must agree to use reliable contraception (e.g., hormonal, barrier, or abstinence) during the study and for at least 90 days after the last dose. Women of childbearing potential must have a negative blood or urine pregnancy test within 7 days prior to the first dose.

  9. Subjects must voluntarily sign the written informed consent form after being informed about the study.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. Received chemotherapy, biologic therapy, targeted therapy, or immunotherapy within 4 weeks prior to first dose; radiotherapy, endocrine therapy, or oral fluoropyrimidines within 2 weeks;traditional Chinese medicine with antitumor indications within 1 week;or nitrosoureas/mitomycin C within 6 weeks.
2. Participation in another investigational drug or therapy trial within 4 weeks prior to first dose.
3. Major surgery (excluding biopsy) or significant trauma within 4 weeks prior to first dose, or scheduled elective surgery during the study.
4. Prior treatment with IL-10-targeted agents.
5. Systemic corticosteroids (prednisone >10 mg/day or equivalent) or immunosuppressants within 14 days prior to first dose, except for: topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids; short-term prophylactic steroids (e.g., to prevent contrast reactions).
6. Immunomodulatory agents (e.g., thymosin, IL-2, interferons) within 14 days prior to first dose.
7. Live or attenuated vaccines within 4 weeks prior to first dose.
8. Prior allogeneic stem cell or organ transplantation.
9. Unresolved adverse events from prior anticancer therapy (excluding alopecia, Grade 2 peripheral neuropathy, or well-controlled hypothyroidism), unless ≤ Grade 1 per CTCAE v5.0.
10. Meningeal metastases, spinal cord compression, or unstable brain metastases requiring steroids or anti-epileptic drugs within 4 weeks before enrollment. Stable brain metastases off steroids/anti-epileptics for ≥4 weeks are allowed.
11. Active infection requiring systemic treatment.
12. Tumor thrombus involving major blood vessels or adjacent organ invasion (e.g., stomach, aorta, trachea) posing high risk of bleeding/perforation, or existing bleeding/perforation/fistula.
13. Known gastrointestinal disorders such as irritable bowel syndrome with symptoms (e.g., chronic nausea, vomiting, diarrhea) or gastric outlet obstruction.
14. History of immunodeficiency, including HIV antibody positivity.
15. Active syphilis, active hepatitis B [HBsAg-positive and HBV DNA >200 IU/mL or above assay's lower limit of detection], or active hepatitis C (HCV antibody positive but HCV RNA below assay limit is allowed). Patients on non-interferon antiviral therapy are eligible.
16. Interstitial lung disease (excluding radiation-induced fibrosis not requiring steroids).
17. Serious cardiovascular or cerebrovascular conditions, including but not limited to:

    * Significant arrhythmia or conduction abnormalities (e.g., Grade II-III AV block requiring intervention)
    * QTcF >470 ms (female) or >450 ms (male)
    * Acute coronary syndrome, heart failure, aortic dissection,stroke, or other Grade ≥3 events within 6 months
    * NYHA class ≥II heart failure or LVEF <50%
    * Uncontrolled hypertension (resting BP ≥160/100 mmHg)
18. Active or recurrent autoimmune disease (e.g., SLE, RA, Crohn's, UC, vasculitis), except for: hypothyroidism requiring hormone replacement or stable type 1 diabetes on insulin.
19. Prior immune-related adverse event (irAE) of Grade ≥3 due to immunotherapy.
20. Clinically uncontrolled third-space or pericardial effusion requiring repeated drainage.
21. Grade ≥3 infusion-related reaction to previous biologic/protein therapy.
22. Known alcohol or substance abuse.
23. Psychiatric illness or poor compliance.
24. Pregnant or breastfeeding women.
25. History of other malignancies within the past 3 years, except for: non- melanoma skin cancer, biopsy-confirmed cervical carcinoma in situ, squamous intraepithelial lesion on Pap test, localized prostate cancer (Gleason <6), or completely resected in situ melanoma. Other low-risk or in-situ cancers may be allowed after sponsor consultation. 26. Other serious systemic diseases or conditions deemed unsuitable by the investigator.

27. Known HER2 positivity, MSI-H/dMMR, or mutations (e.g., KRAS) for which approved targeted therapies are available per guidelines.

28. Grade IV myelosuppression related to prior antitumor therapy. 29. Primary or secondary platelet count decreased or platelet-destructive diseases (e.g., Fanconi anemia, congenital platelet count decreased without megakaryocytes, May-Hegglin anomaly, aplastic anemia, bone marrow infiltration, radiation to bone marrow, megakaryocytic hypoplasia, ITP). 30. Arterial or venous thrombotic events within 6 months, including stroke (TIA, cerebral hemorrhage, infarction), DVT, or pulmonary embolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
MTD/RP2D | up to study completion,approximately 24 months
  MTD is determined based on the occurrence of DLTs. In this study, MTD is defined as the dose level at which 0/3 or 1/6 subjects experience a DLT, and at the next higher dose level, at least 2/3 or 2/6 subjects experience a DLT.
DLT occurrence and frequency (dose escalation phase) | The first period of LB4330 treatment (28 days for the first subject in the first dose group, 21 days for the rest subjects. If the administration is delayed, the DLT evaluation period should be extended to 7 days after the third administration)
  The DLT evaluation period is the first cycle of LB4330 treatment (28 days for the first subject in the first dose cohort, and 21 days for all other subjects. If a dosing delay occurs, the DLT evaluation period should be extended accordingly to 7 days after the third administration).
AE, SAE occurrence and frequency (according to NCI CTCAE 5.0) | up to 90 days following last dose
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Serum PK parameters | Up to finished treatment
  AUC0-t and so on.
Pharmacodynamic index | through study completion, an average of 8 months.
  Pharmacodynamic index: percentage of monocytes
Immunogenicity | up to 90 days following last dose
  Immunogenicity index: positive rate, titer and duration of ADA; neutralizing antibody (NAb) analysis will be conducted if necessary.
Overall response rate (ORR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST).
Disease control rate (DCR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST).
Progression-free survival (PFS) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST).
Duration of response (DOR) | through study completion, an average of 8 months.
  Evaluation Criteria in Solid Tumors (RECIST) v 1.1 and Immunotherapeutics Response Evaluation Criteria in Solid Tumors (iRECIST).
OS | through study completion，an average of 1 year
  Total survival period (OS): It is defined as the time from the start of using the study drug to the death due to any reason.
Biomarker | through study completion, an average of 8 months.
  Biomarker: relationship between Claudin 18.2 expression level in tumor tissue and clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, Doctor, Principal Investigator — Fudan University; Jian Zhang, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China